CLINICAL TRIAL: NCT05006105
Title: Early Detection of Atrial Fibrillation Using Mobile Technology in Cryptogenic Stroke Patients - REMOTE Study
Brief Title: Early Detection of Atrial Fibrillation Using Mobile Technology in Cryptogenic Stroke Patients
Acronym: REMOTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziekenhuis Oost-Limburg (Other)
Collaborators: Hasselt University (Other); Jessa Hospital (Other)
Responsible Party: Principal Investigator, David Verhaert, MD, Dr., Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CTU2019106
Record Dates: First submitted 2021-07-13; First posted 2021-08-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Cryptogenic Stroke; Atrial Fibrillation
Keywords: Mobile health; Prolonged cardiac monitoring; Photoplethysmography
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation | interventions — Electrocardiography, Ambulatory; Blood Pressure Monitors

STUDY DESIGN:
Intervention Model Description: Group 1 uses PPG-based mHealth with a smartphone; two times a day, a spot-check measurement is taken; and in case of symptoms, additional measurements can be taken.
  Group 2 uses PPG-based mHealth with a smartwatch, this results in semi-continuous measurements that are performed automatically.
Who Masked: Participant, Care Provider
Masking Description: The participant and care provider are not blinded for which mHealth method is used (smartphone or smartwatch), but are blinded for the mHealth results (i.e., AF detection) during the monitoring period with the mHealth application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPG-based mHealth on smartphone (Experimental): Participants used PPG-based mHealth on a smartphone for 6 months. Participants were asked to perform two spot-check measurements and additional measurements in case of symptoms. The use of PPG-based mHealth on a smartphone was initiated on the day of insertable loop recorder insertion.
  Interventions: Device: seven-day ECG Holter; Device: 24-hour blood pressure monitor; Other: Questionnaire: vision of mHealth; Other: Questionnaire: user experience & feeling of safety; Device: Insertable loop recorder
- PPG-based mHealth on smartwatch (Experimental): Participants used PPG-based mHealth on a smartwatch for 6 months. Participants were asked to wear the smartwatch continuously (except during battery charging). The use of PPG-based mHealth on a smartwatch was initiated on the day of insertable loop recorder insertion.
  Interventions: Device: seven-day ECG Holter; Device: 24-hour blood pressure monitor; Other: Questionnaire: vision of mHealth; Other: Questionnaire: user experience & feeling of safety; Device: Insertable loop recorder

INTERVENTIONS:
Device: seven-day ECG Holter — Participants receive a seven-day ECG Holter after hospital discharge.
Device: 24-hour blood pressure monitor — Participants receive a 24-hour blood pressure monitor, approximately four weeks after hospital discharge.
Other: Questionnaire: vision of mHealth — Participants receive a questionnaire concerning their vision of mHealth, approximately four weeks after hospital discharge.
Other: Questionnaire: user experience & feeling of safety — Participants receive a questionnaire concerning their user experience and feeling of safety of using mHealth, after using mHealth for six months.
Device: Insertable loop recorder — Participants receive an insertable loop recorder, approximately six weeks after hospital discharge.

SUMMARY:
The purpose of this study is to demonstrate the added value of mobile health (mHealth) to detect atrial fibrillation (AF) early in the care path of cryptogenic stroke and transient ischemic attack (TIA) patients.

DETAILED DESCRIPTION:
The use of photoplethysmography (PPG)-based mHealth (with smartphone and smartwatch) is compared to the guideline-recommended insertable loop recorders (ILR) in the detection of AF in cryptogenic stroke or TIA patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cryptogenic ischemic stroke or TIA
* The patient or its legal representative is willing to sign the informed consent

Exclusion Criteria:

* History of AF or atrial flutter
* Life expectancy of less than one year
* Not qualified for ILR insertion
* Indication or contraindication for permanent oral anticoagulants (OAC) at enrolment
* Untreated hyperthyroidism
* Myocardial infarction or coronary bypass grafting less than one month before the stroke onset
* Presence of patent foramen ovale (PFO) and it is or was an indication to start OAC according to the European Stroke Organization guidelines
* Inclusion in another clinical trial that will affect the objectives of this study
* Not able to understand the Dutch language
* Patient or partner not in possession of a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
AF detection with mHealth versus ILR - Percentage | After 6 months of having an ILR inserted and using mHealth.
  Percentage of patients with AF detected

SECONDARY OUTCOMES:
AF detection with ILR - Percentage | After 12 months of having an ILR inserted.
  Percentage of patients with AF detected
AF detection with mHealth versus ILR - Time to first AF detection | Baseline until end of study (after 12 months of having an ILR inserted).
  Time to first AF detection
AF detection with mHealth versus ILR - Frequency | Baseline until end of study (after 12 months of having an ILR inserted).
  Frequency of AF episodes
AF detection with mHealth versus ILR - Duration | Baseline until end of study (after 12 months of having an ILR inserted).
  Duration of AF episodes
User experience and feeling of safety questionnaire | After 6 months of having an ILR inserted and using mHealth.
  Questionnaire with a 7 point Likert scale
Correlation between baseline characteristics and AF detection | Baseline until end of study (after 12 months of having an ILR inserted).
  Baseline characteristics include comorbidities, results of standard of care in-hospital stroke examinations and scores, relevant in-hospital therapy
Correlation between follow-up characteristics and AF detection | Baseline until end of study (after 12 months of having an ILR inserted).
  Follow-up characteristics include changes in therapy, number of relevant readmissions, mortality and healthcare-related costs

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Ziekenhuist Oost-Limburg, Genk, Limburg
  - Jessa Hospital, Hasselt, Limburg